CLINICAL TRIAL: NCT02807259
Title: Evaluation of Samvedana Plus: An Intervention With Female Sex Workers (FSWs) and Their Intimate Partners to Reduce Partner Violence and Increase Consistent Condom Use Within Intimate Relationships
Brief Title: Reducing Vulnerability in the Intimate Partnerships of Female Sex Workers Sex Workers
Acronym: SamPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karnataka Health Promotion Trust (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SamPlus01
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Violence; Sexual Behaviour; HIV
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-level intervention (Experimental): This is a cluster-randomised controlled trial design. The unit of randomisation is village.
  Interventions: Behavioral: Multi-level intervention
- Control (Other): The intervention will rolled out to all participating villages after 24 months.
  Interventions: Behavioral: Multi-level intervention

INTERVENTIONS:
Behavioral: Multi-level intervention — At the individual level, the intervention will focus on: (i) structured reflection groups for FSWs to enhance self-esteem, encourage critical reflection around gender norms and violence, and build individual and collective efficacy; (ii) separate sessions for intimate partners to discuss issues around violence and condom use as well as gender, equity, respect and responsibility; (iii) skills building around female condoms (iv) access to individual and couples-based counselling. At the community level, the intervention will focus on: (i) strengthening the supportive crisis management systems so that they are able to address 'domestic' as well as 'work-place' violence among FSWs and (ii) building an environment that encourages action against violence from intimate partners by training male champions and developing folk media troops to generate discussion around gender, masculinity, violence and HIV risk behaviours.

SUMMARY:
Female sex workers (FSWs) frequently experience violence from their intimate partners (non-paying lovers), which compromises their health and increases their the risk of infection with HIV or other sexually transmitted infections. Samdevena Plus is a complex multi-level intervention that works with FSWs, their intimate partners, the sex worker community and the general population. The intervention aims to reduce partner violence and increase consistent condom use within these relationships.

The intervention consists of: (i) couples counselling sessions between FSWs and their intimate partners; (ii) separate group work among FSWs and intimate partners to increase self-esteem and encourage reflection about violence; (iii) strengthening supportive crisis management systems that address domestic and sex worker violence; (iv) training male 'champions' to encourage action against violence; and (v) training media to promote informed discussions about violence and HIV risk.The program involves changing perceptions on acceptability of physical violence as a form of discipline, challenging assumptions that give men authority over women, and working with men and women to encourage new relationship models based on equality and respect. The intervention will reach 800 FSWs and their intimate partners living in 47 villages in north Karnataka, India. The evaluation uses a cluster-randomized control trial design that introduces the intervention into half of villages for the first 24 months and the remaining half receive the intervention thereafter. The primary outcomes of the trial are: the proportion of FSWs who report: i) consistent condom use in their intimate relationship; and ii) experiencing partner violence within the past 6 months.

DETAILED DESCRIPTION:
Female sex workers (FSWs) are at increased risk of HIV and sexually transmitted infections (STI) compared to women in the general population, and frequently experience violence in their working and domestic lives from a variety of perpetrators, which can enhance this risk. While progress has been made in addressing violence by police and clients, little work has been done to understand and prevent violence by intimate partners (IPs) among FSW populations.

Samvedana Plus is a multi-level intervention programme that works with FSWs, their IPs, the sex worker community, and the general population, and aims to reduce violence and increase consistent condom use within these 'intimate' relationships. The programme involves shifting norms around the acceptability of beating as a form of discipline, challenging gender roles that give men authority over women, and working with men and women to encourage new relationship models based on gender equity and respect. The programme will aim to cover 800 FSWs and their IPs living in 47 villages in Bagalkot district, northern Karnataka. The study is designed to assess three primary outcomes: the proportion of FSWs who report: (i) any physical or sexual partner violence; (ii) severe/moderate physical or sexual partner violence in the last 6 months; and iii) consistent condom use in their intimate relationship. The evaluation will employ a cluster-randomised controlled trial design, with 50% of the village clusters (n=24) randomly selected to receive the intervention for the first 24 months and the remaining 50% (n=23) receiving the intervention thereafter. Statisticians will be blinded to treatment arm allocation. The evaluation will use an adjusted, individual-level intention to treat analysis, comparing outcomes in intervention and control villages at endline (24 months) using a mixed effects logistic model. We will adjust for confounders in two ways: i) outcome variables are adjusted for at a cluster level using the mean baseline summaries; ii) other variables will be adjusted for an at an individual level using endline data. We will include all women survey at endline. We will also report cluster-level summaries by trial arm for each primary and secondary outcome to double check our analyses. The evaluation design will involve quantitative and qualitative assessments with (i) all FSWs who report an IP (ii) IPs; and process/ implementation monitoring.

This is an innovative intervention programme that aims to address violence by IPs as part of HIV prevention programming with FSWs. Reducing violence is expected to reduce vulnerability to HIV acquisition, and help women to work and live without fear of violence.

ELIGIBILITY:
Inclusion Criteria:

* Female Sex Workers who engage in commercial sex and who currently have an intimate partner or have had an intimate partner in the last 6 months, living in any of the 47 villages.

Exclusion Criteria:

* Female sex workers aged younger than 18 years, who do not have an intimate partner or have not had one in the last 6 months, or who live outside of the villages.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Heise, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Karnataka Health Promotion Trust, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised and made available for secondary analyses on request, following publication of trial findings.

REFERENCES:
- [Derived] Javalkar P, Platt L, Prakash R, Beattie TS, Collumbien M, Gafos M, Ramanaik S, Davey C, Jewkes R, Watts C, Bhattacharjee P, Thalinja R, Dl K, Isac S, Heise L. Effectiveness of a multilevel intervention to reduce violence and increase condom use in intimate partnerships among female sex workers: cluster randomised controlled trial in Karnataka, India. BMJ Glob Health. 2019 Nov 6;4(6):e001546. doi: 10.1136/bmjgh-2019-001546. eCollection 2019. PMID 31798984
- [Derived] Javalkar P, Platt L, Prakash R, Beattie T, Bhattacharjee P, Thalinja R, L KD, Sangha CATM, Ramanaik S, Collumbien M, Davey C, Moses S, Jewkes R, Isac S, Heise L. What determines violence among female sex workers in an intimate partner relationship? Findings from North Karnataka, south India. BMC Public Health. 2019 Mar 29;19(1):350. doi: 10.1186/s12889-019-6673-9. PMID 30922283
- [Derived] Beattie TS, Isac S, Bhattacharjee P, Javalkar P, Davey C, Raghavendra T, Nair S, Ramanaik S, Kavitha DL, Blanchard JF, Watts C, Collumbien M, Moses S, Heise L. Reducing violence and increasing condom use in the intimate partnerships of female sex workers: study protocol for Samvedana Plus, a cluster randomised controlled trial in Karnataka state, south India. BMC Public Health. 2016 Jul 29;16:660. doi: 10.1186/s12889-016-3356-7. PMID 27473180

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: villages
Groups:
- Samvedana Plus Multi-level Intervention: In brief, the programme, informed by prior participatory research, worked with individuals, couples, and at a community level to change the acceptability of IPV as a form of discipline, to challenge assumptions that give men authority over women, and to encourage new relationship models based on equality and respect. The intervention, implemented between April 2015 and September 2017, lasted 27 months (Box 1). It was led by a local community-based organisation (CBO) sex worker collective Chaitanya AIDS Tadegattuva Mahila Sangha (CATMS) in collaboration with the Karnataka Health Promotion Trust (KHPT). The CBO was responsible for identifying sex workers and IPs to take part in the intervention; with support from KHPT they trained outreach workers to facilitate 12 reflection sessions and provide counselling, training male champions; and building alliances with other networks to address violence against sex workers.
- Wait List Control: Villages in the control arm continued to receive standard HIV programming (including condom distribution and HIV prevention information via peer educators) and at month 24 began to receive the intervention.
Period: Baseline (3 Months)
Arm/Group | Samvedana Plus Multi-level Intervention | Wait List Control
Started | 405; 24 villages | 404; 23 villages
Completed | 328; 24 villages | 292; 23 villages
Not Completed | 77; 0 villages | 112; 0 villages
Not completed — migration, refusal, not available | 77 | 112
Period: Midline (3 Months)
Arm/Group | Samvedana Plus Multi-level Intervention | Wait List Control
Started | 352; 24 villages | 223; 23 villages
Completed | 322; 24 villages | 189; 23 villages
Not Completed | 30; 0 villages | 34; 0 villages
Not completed — migration, refusal, not available | 30 | 34
Period: Endline (3 Months)
Arm/Group | Samvedana Plus Multi-level Intervention | Wait List Control
Started | 323; 24 villages | 346; 23 villages
Completed | 288; 24 villages | 259; 23 villages
Not Completed | 35; 0 villages | 87; 0 villages
Not completed — migration, refusal, not available | 35 | 87

BASELINE CHARACTERISTICS:
Groups:
- Samvedana Plus Multi-level Intervention: Multi-level intervention working with sex workers, their intimate partners and communities to reduce intimate partner violence (IPV) and increase condom use
- Wait-list Control: Wait list control.
- Total: Total of all reporting groups
Arm/Group | Samvedana Plus Multi-level Intervention | Wait-list Control | Total
Number analyzed (Participants) | 328 | 292 | 620
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (7.0) | 35.2 (7.6) | 34.5 (7.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 328 | 292 | 620
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 328 | 292 | 620
Cluster level mean of any IPV (physical or sexual violence) in past 6 months [Mean (Standard Deviation); unit: Mean percentage of participants] | 31.4 (22.4) | 45.0 (24.6) | 38.0 (24.2)
Cluster level mean of severe IPV (physical and/or sexual violence) in the past 6 months [Mean (Standard Deviation); unit: Mean percentage of participants] | 23.7 (21.1) | 33.8 (23.9) | 28.6 (22.8)
Cluster level mean of consistent condom use within the past 30 days [Mean (Standard Deviation); unit: Mean percentage of participants] | 38.9 (31.7) | 46.0 (23.2) | 42.4 (27.8)
Cluster level mean of acceptance IPV from their intimate partners [Mean (Standard Deviation); unit: Mean percentage of participants] | 59.2 (22.8) | 55.1 (21.5) | 57.2 (22.1)
Cluster level mean of disclosure of IPV [Mean (Standard Deviation); unit: Mean percentage of participants] | 46.3 (32.5) | 52.1 (28.9) | 49.1 (30.6)
Cluster level mean of knowledge of self-protection strategies against IPV [Mean (Standard Deviation); unit: Mean percentage of participants] | 6.2 (7.6) | 7.0 (9.0) | 6.6 (8.2)
Cluster level mean of self-efficacy to negotiate condom use with intimate partner [Mean (Standard Deviation); unit: Mean percentage of participants] | 19.9 (17.9) | 20.0 (21.3) | 20.0 (19.4)
Cluster level mean of solidarity around issues of IPV [Mean (Standard Deviation); unit: Mean percentage of participants] | 15.0 (20.0) | 22.0 (20.3) | 18.4 (20.2)
Cluster level mean of village population size [Mean (Standard Deviation); unit: Number of residents] | 4121 (2694.3) | 3755 (2350.1) | 3942 (2511.0)
Cluster level mean of sex work population size [Mean (Standard Deviation); unit: Number of sex workers] | 17.2 (13.7) | 16.9 (14.8) | 17.0 (14.1)

OUTCOME MEASURES:

1. Primary Outcome: Intimate Partner Violence
Description: Proportion of FSWs who report experiencing any intimate partner violence in the last 6 months
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Samvedana Plus Multi-level Intervention | Wait List Control
Number analyzed (Participants) | 288 | 259
Participants | 26 | 21
Statistical Analysis 1: Comparison: Samvedana Plus Multi-level Intervention vs Wait List Control; Power calculations were conducted assuming an IPV prevalence (past 12 months) of 47% and consistent condom use (past 12 months) of 38% based on initial assessments. The power calculation was performed by analysing simulated data from 800 women, distributed across clusters using empirical data with a range in variance across cluster-level proportions of IPV (15% to 25% of the total variation) and a narrow range of effect sizes (risk ratio= 0.75-0.80); Test type: Equivalence — Power calculations did not account for stratification used in the randomisation or include adjustment for baseline levels of the outcome, since the correlation over time was not known. Results suggested that the trial had >80% power to detect a risk ratio of 0.77, if the coefficient of between-cluster variation was between 0.15 and 0.25; p = 0.298, Mixed Models Analysis; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.71 to 3.01]

2. Primary Outcome: Severe Intimate Partner Violence
Description: Proportion of sex workers experienced severe physical and/or sexual violence from intimate partners in the past 6 months
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Groups:
- Wait-list Control: Peer educators, HIV counselling, condom distribution. The intervention will rolled out to all participating villages after 24 months.
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 25 | 18
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.378, Mixed Models Analysis; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.68 to 2.81]

3. Primary Outcome: Condom Use
Description: Proportion of sex workers who report consistent condom use in their intimate relationship in the last 30 days
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 165 | 162
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.748, Mixed Models Analysis; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.58 to 1.47]

4. Secondary Outcome: Changes in Acceptance of Violence
Description: Change in the proportion of FSWs who report violent actions from intimate partners to be unacceptable
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 193 | 188
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.025, Mixed Models Analysis; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.4 to 0.94]

5. Secondary Outcome: Change in Disclosure of Violence From Intimate Partners
Description: Change in proportion of FSWs who are willing to disclose incidences of violence by their intimate partner
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 21 | 15
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.372, Mixed Models Analysis; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.42 to 10.26]

6. Secondary Outcome: Changes in Self-efficacy
Description: Proportion of FSWs who report ability to negotiate condom use and HIV/STI testing by their IP
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 170 | 163
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.845, Mixed Models Analysis; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.61 to 1.50]

7. Secondary Outcome: Changes in Solidarity Among FSWs Around Violence
Description: Change in proportion of FSWs who support their peers to reduce incidences of violence among FSWs
Time Frame: 27 months after implementing the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-level Intervention | Wait-list Control
Number analyzed (Participants) | 288 | 259
Participants | 112 | 81
Statistical Analysis 1: Comparison: Multi-level Intervention vs Wait-list Control; Test type: Other; p = 0.042, Mixed Models Analysis; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.02 to 2.82]

ADVERSE EVENTS:
Time Frame: Data on adverse events were monitored for the duration of the intervention implementation (27 months).
Description: A community advisory board of sex workers was set up to inform all aspects of study design, implementation and consent procedures, to ensure it was acceptable to the community and to help monitor any adverse events (defined as a report of sexual/physical violence). Outreach workers collected reports of violence during regular sessions with sex workers, completing a report when incidents occurred. These reports were monitored and reported to the Crisis Management Committee.
Groups:
- Control: Peer educators, HIV counselling, condom distribution. The intervention will rolled out to all participating villages after 24 months.
Arm/Group | Multi-level Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/292
Serious Adverse Events (participants affected / at risk) | 0/328 | 0/292
Other Adverse Events (participants affected / at risk) | 0/328 | 0/292

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02807259/SAP_000.pdf
  • Study Protocol (2014-07-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT02807259/Prot_001.pdf